CLINICAL TRIAL: NCT04298918
Title: A Phase lb/ll, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Venetoclax in Combination With Trastuzumab Emtansine in Patients With Previously Treated HER2-Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study Evaluating the Safety and Efficacy of Venetoclax in Combination With Trastuzumab Emtansine in Patients With Previously Treated HER2-Positive Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision to discontinue the study based on broader development and strategic prioritisation. The Sponsor concludes there is no benefit-risk impact on the CO41863 study.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO41863; 2019-004200-35 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — venetoclax; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Phase (Experimental): Participants received venetoclax in combination with a fixed dose of trastuzumab emtansine.
  Interventions: Drug: Venetoclax; Drug: Trastuzumab emtansine
- Dose Expansion Phase (Experimental): Participants were to receive venetoclax at the Phase II Recommended Dose (RP2D) in combination with trastuzumab emtansine.
  Interventions: Drug: Venetoclax; Drug: Trastuzumab emtansine
- Randomized Phase II Arm 1 (Experimental): Participants were to receive trastuzumab emtansine + placebo.
  Interventions: Drug: Placebo; Drug: Trastuzumab emtansine
- Randomized Phase II Arm 2 (Experimental): Participants were to receive trastuzumab emtansine + venetoclax.
  Interventions: Drug: Venetoclax; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Placebo — Participants will receive oral placebo in combination with trastuzumab emtansine.
  Arms: Randomized Phase II Arm 1
Drug: Venetoclax — Participants will receive oral venetoclax.
  Other Names: Venclexta
  Arms: Dose Escalation Phase; Dose Expansion Phase; Randomized Phase II Arm 2
Drug: Trastuzumab emtansine — Participants will receive intravenous (IV) trastuzumab emtansine.
  Other Names: Kadcyla

SUMMARY:
This two-part study is composed of two stages: a Phase Ib stage consisting of a dose-escalation phase and an expansion phase; and a Phase II, randomized, placebo-controlled, double-blind, multicenter stage. The Phase Ib stage will assess the safety and tolerability, determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D), and evaluate the preliminary efficacy of trastuzumab emtansine in combination with venetoclax in participants with previously treated human epidermal growth factor receptor 2 (HER2) positive unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (MBC). Additional patients may be enrolled in an expansion phase to evaluate the safety, tolerability, and efficacy of trastuzumab emtansine in combination with venetoclax at RP2D in patients with previously treated HER2-positive LABC or MBC who have previously received either trastuzumab emtansine or trastuzumab deruxtecan (DS-8201a). The Phase II randomized stage will evaluate the safety, efficacy, tolerability, and pharmacokinetics of trastuzumab emtansine in combination with venetoclax at RP2D compared with trastuzumab emtansine plus placebo in participants with previously treated HER2-positive LABC or MBC who have not received prior trastuzumab emtansine therapy, either alone or in combination with other anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed invasive metastatic breast cancer (MBC) or locally advanced breast cancer (LABC) that is incurable, unresectable, and previously treated with multimodality therapy
* Measurable disease that is evaluable per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Willing to provide tumor biopsy sample at the time of screening
* Local histological or cytological confirmation of estrogen receptor (ER) and/or progesterone receptor status as defined by using immunohistochemistry (IHC) per American Society of Clinical Oncology/College of American Pathologists criteria
* Percentage of ER and/or progesterone receptor positivity, if available
* Willing to provide blood samples at the time of screening, on-study, and at progression for exploratory research on biomarkers
* HER2-positive BC as defined by an IHC score of 3+ or gene amplified by in situ hybridization (ISH) as defined by a ratio of >/= 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies
* Adequate hematologic and end-organ function
* Screening left ventricular ejection fraction (LVEF) >/= 50% on echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
* Negative HIV test, hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax or 7 months after the last dose of trastuzumab emtansine
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm during the treatment period and for at least 30 days after the last dose of venetoclax or 7 months after the last dose of trastuzumab emtansine

Inclusion Criteria for Expansion Phase Only

In addition to the general inclusion criteria, participants in the expansion phase must also meet the following criteria for study entry:

* Trastuzumab emtansine experienced cohort: Disease progression during or after trastuzumab emtasine in the advanced/metastatic setting or disease recurrence in the neoadjuvant/adjuvant setting; At least 50% of participants in the expansion cohort must have a tumor that is Bcl-2 high (defined as >50% of tumor cells stained with an intensity of immunohistochemistry (IHC) 2+ or 3+)
* Trastuzumab deruxtacan (DS-8201a) experienced cohort: Disease progression during or after trastuzumab deruxtecan in the advanced/metastatic setting; Prior trastuzumab emtansine in any setting is allowed; At least 50% of participants in the expansion cohort must have a tumor that is Bcl-2 high

Exclusion criteria

* Receipt of any anticancer drug/biologic or investigational treatment 21 days prior to Cycle 1, Day 1 except hormone therapy, which can be given up to 7 days prior to Cycle 1, Day 1
* Radiation therapy within 2 weeks prior to Cycle 1, Day 1
* History of exposure to the following cumulative doses of anthracyclines as specified: Doxorubicin >500 mg/m2; Liposomal doxorubicin >500 mg/m2; Epirubucin >720 mg/m2; Mitoxantrone >120 mg/m2; Idarubicin >90 mg/m2. If another anthracycline or more than one anthracycline has been used, then the cumulative dose must not exceed the equivalent of 500 mg/m2 doxorubicin.
* History of other malignancy within the previous 5 years
* Cardiopulmonary dysfunction
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, autoimmune hepatic disorders, sclerosis cholangitis, or active infection with HBV or HCV)
* Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* Known HIV infection or human T-cell leukemia virus 1 infection
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization
* Known central nervous system (CNS) disease
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Current Grade >/= 3 peripheral neuropathy
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies, excipients of any drugs formulated in polysorbate 80 or 20 or fusion proteins
* Prior allogeneic stem cell or solid organ transplantation
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 30 days after the last dose of venetoclax or 7 months after the last dose of trastuzumab emtansine after the final dose of study treatment, whichever is later
* Consumption of grapefruit, grapefruit products, Seville oranges, or starfruit within 3 days before anticipated first dose of study drug until the last dose of study drug
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* History of active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) requiring specific medication in the 12 months prior to randomization, or active and uncontrolled bowel inflammation (e.g., diverticulitis) at time of randomization
* Inability or unwillingness to swallow a large number of tablets
* Known hypersensitivity to venetoclax or trastuzumab emtansine or to any of their excipients
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Other medical or psychiatric conditions that, in the opinion of the investigator, may interfere with the patient's participation in the study
* Blood transfusions if performed within 2 weeks prior to screening

Exclusion Criteria for Randomized Phase II Stage

In addition to the general exclusion criteria, participants in the randomized Phase II stage who meet the following criteria will be excluded:

* Prior treatment with trastuzumab emtansine in any setting (neoadjuvant/adjuvant or advanced/metastatic setting)
* Prior treatment with venetoclax in any setting
* Prior treatment with anti-HER2 antibody drug conjugates (e.g. trastuzumab deruxtecan [DS-8201a]), margetuximab, pyrotinib, or tucatinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Peter MacCallum Cancer Center, East Melbourne, Victoria, Australia
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | Dose Escalation Phase | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: Participants]
Race/Ethnicity, Customized [unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Number of Participants With Adverse Events
Description: The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline up until 28 days after the last dose of study drug or until initiation of new systemic anti-cancer therapy, whichever occurs first (up to a maximum of 20 weeks).
Population: as for baseline characteristics
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 0

2. Primary Outcome: Expansion Phase: Objective Response Rate (ORR)
Description: as for outcome 1
Time Frame: Up to 30 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 0

3. Primary Outcome: Phase II: ORR
Description: as for outcome 1
Time Frame: Up to 30 months
Population: as for baseline characteristics
Arm/Group | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Phase II: Progression-Free Survival (PFS)
Description: as for outcome 1
Time Frame: Up to 30 months
Population: as for baseline characteristics
Arm/Group | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: All Phases: Plasma Concentration of Venetoclax
Description: as for outcome 1
Time Frame: At pre-defined time points from Cycle 1 Day 8 and/or Cycle 2 Day 1 through Cycle 4 Day 1 (cycle = 21 days)
Population: as for baseline characteristics
Arm/Group | Dose Escalation Phase | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Phase II: Serum Concentration of Trastuzumab Emtansine
Description: as for outcome 1
Time Frame: At pre-defined time points from Cycle 1 Day 1 through Cycle 4 Day 1 (cycle = 21 days)
Population: as for baseline characteristics
Arm/Group | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Expansion Phase and Phase II: Number of Participants With Adverse Events
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for baseline characteristics
Arm/Group | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Expansion Phase and Phase II: Duration of Response (DOR)
Description: as for outcome 1
Time Frame: Up to 30 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Phase II: Overall Survival (OS)
Description: as for outcome 1
Time Frame: Randomization to death from any cause (up to 30 months)
Population: as for baseline characteristics
Arm/Group | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase II: Number of Participants With Anti-Drug Antibodies (ADAs) to Trastuzumab Emtansine
Description: as for outcome 1
Time Frame: Up to 30 months
Population: as for baseline characteristics
Arm/Group | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Dose Escalation Phase | Dose Expansion Phase | Randomized Phase II Arm 1 | Randomized Phase II Arm 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT04298918/Prot_SAP_000.pdf